CLINICAL TRIAL: NCT01142245
Title: Phase 3 Study of Effect of Intravenous and Oral Esomeprazole in Prevention of Recurrent Bleeding From Peptic Ulcers After Endoscopic Therapy (IOE Study)
Brief Title: Effect of IV and Oral Esomeprazole in Prevention of Recurrent Bleeding From Peptic Ulcers After Endoscopic Therapy
Acronym: IOE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IOE
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Peptic Ulcer; Bleeding
Keywords: ulcer bleeding; endoscopic therapy
MeSH Terms: conditions — Peptic Ulcer; Hemorrhage | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral esomeprazole (Active Comparator): * Esomeprazole placebo IV loading bolus
  * Esomeprazole placebo intravenous infusion for 72 hours
  * Oral Esomeprazole: 80 mg/Day on Day 1, 2 and Day 3, and the drug will be given as 40 mg q12h.
  Interventions: Drug: Oral esomeprazole
- Intravenous Esomeprazole (Active Comparator): Esomeprazole IV loading bolus 80mg
  • Esomeprazole intravenous infusion 8mg/hr for 72 hours
  Interventions: Drug: Intravenous Esomeprazole

INTERVENTIONS:
Drug: Oral esomeprazole — • Oral Esomeprazole 40mg on Day 1, 2 and Day 3 q12h
  Other Names: oral; nexium
  Arms: oral esomeprazole
Drug: Intravenous Esomeprazole — Esomeprazole IV 80mg loading bolus
  * Esomeprazole intravenous infusion 8mg/hr for 72 hours
  Other Names: IV; nexium
  Arms: Intravenous Esomeprazole

SUMMARY:
The investigators previously showed that the use of a high-dose intravenous PPI regimen after endoscopic control of bleeding from peptic ulcers reduced rate of recurrent bleeding, decreased the need for endoscopic and surgical interventions and in general improved patients' outcomes. A trend towards reduced mortality associated with the use of high-dose intravenous PPI was also observed. Recent clinical trials from Asia have provided evidence that high-dose oral PPIs are associated with a reduction in rebleeding. Current meta-analysis suggests that both high dose (intravenous) and low dose (oral) PPIs effectively reduce rebleeding vs placebo. However, there has been no clinical study to compare IV infusion to oral PPI in this patient population.

The purpose of this clinical study is to compare the efficacy and safety of intravenous and oral Esomeprazole in patients with peptic ulcer hemorrhage who are at risk for recurrent bleeding. The investigators hypothesize that using IV infusion is superior to oral PPI.

DETAILED DESCRIPTION:
The investigators previously showed that the use of a high-dose intravenous PPI regimen after endoscopic control of bleeding from peptic ulcers reduced rate of recurrent bleeding, decreased the need for endoscopic and surgical interventions and in general improved patients' outcomes. A trend towards reduced mortality associated with the use of high-dose intravenous PPI was also observed. Recent clinical trials from Asia have provided evidence that high-dose oral PPIs are associated with a reduction in rebleeding. Current meta-analysis suggests that both high dose (intravenous) and low dose (oral) PPIs effectively reduce rebleeding vs placebo. However, there has been no clinical study to compare IV infusion to oral PPI in this patient population.

Endoscopic stigmata in bleeding peptic ulcers are prognostic and allow risk stratification. Patients with a clean ulcer base have a < 5% risk of rebleeding; this increases progressively with a flat spot, adherent clot, non-bleeding visible vessel and active bleeding (55%). Early endoscopy in patients with bleeding peptic ulcers selects the high risk ulcers for therapy and evaluation of adjuvant PPI use.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Confirmed ulcer bleeding with Forrest Ia, Ib, IIa, IIb
* Endoscopic hemostasis achieved
* Informed consent obtained

Exclusion Criteria:

* No consent
* Forrest II c, III (clear ulcer base/flat spot and no active bleeding, i.e., minimal risk for rebleeding)
* Unsuccessful endoscopic treatment (i.e., injection and/or thermal coagulation for the initial bleeding) or severe bleeding that immediate surgery is indicated
* Moribund patients in whom active treatment of any form is not considered.
* Polytrauma, severe injury, unconsciousness, burns, or need for continuous artificial ventilation
* Upper GI malignancy or disseminated malignant disease
* Esophageal varices
* A Mallory-Weiss lesion
* Phenytoin or theophylline treatment
* Uses of PPI or H2RAs within 3 days of admission, including uses at Emergency Department N.B. Usage of aspirin or NSAID is not an exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2008-01; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Rate of clinical rebleeding within 30 day of endoscopic therapy | 30 days
  Definition of clinical rebleeding
  1. Recurrent hematemesis
  2. fresh melena after normal stool
  3. Hypotension SBP<90 or tachycardia >110 AND fresh melena
  4. Decrease in Hb >2g/dL (or Hct > 10%) during any 24 h or an increas in Hb <1 g/dL (or Hct <3%) despite ≥4 units of blood has been transfused during any 48h

SECONDARY OUTCOMES:
Un-scheduled further endoscopic therapy | 30 days
  * Un-scheduled further endoscopic therapy
  * Need for surgery (i.e., operation rate)
  * Duration of hospitalization
  * Blood transfusion
Need for surgery | 30 days
Duration of hospitalization | 30 days
Blood transfusion | 30 days
mortality | 30 days
need of surgery | 30 days
un-scheduled further endoscopic therapy | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Francis K Chan, MD, Principal Investigator — CUHK
Locations (2):
- China (2):
  - Endoscopy Centre, Hong Kong
  - Endoscopy Center in Prince of Wales Hospital, Hong Kong (sar)